CLINICAL TRIAL: NCT00506753
Title: Prison Study: Motivation and Skills for THC/ETOH+ Teens in Jail
Brief Title: Motivation and Skills for Delta-9-tetrahydrocannabinol/Ethanol (THC/ETOH+) Teens in Jail
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lynda Stein, Ph.D., Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA018851-02; R01DA018851 (NIH); NCT00249028 (obsolete NCT alias)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Drinking; Marijuana Smoking
Keywords: substance abuse
MeSH Terms: conditions — Alcohol Drinking; Marijuana Smoking; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy; Relaxation Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MI/CBT (Experimental): Motivational Interviewing followed by Cognitive Behavior Therapy
  Interventions: Behavioral: MI/CBT
- RT/TU (Experimental): Relaxation Training followed by Treatment as Usual
  Interventions: Behavioral: RT/SU

INTERVENTIONS:
Behavioral: MI/CBT — Motivational Interviewing followed by Cognitive Behavior Therapy
  Other Names: Motivation Interviewing,Cognitive Behavior Therapy
  Arms: MI/CBT
Behavioral: RT/SU — Relaxation Training followed by Treatment as Usual
  Other Names: Relaxation Training, Treatment as Usual
  Arms: RT/TU

SUMMARY:
This study will focus on treating substance abusing incarcerated teens using individually administered Motivational Interviewing (MI) followed by group Cognitive Behavior Therapy (CBT). The control group receives individualized Relaxation Training (RT) followed by group Treatment as Usual (TU). Currently, there is little research regarding effective group treatments for incarcerated teens and this study will address this gap in our knowledge base. We seek to reduce substance use and associated risky behaviors post-release (including driving under the influence, risky sexual behaviors, etc.)

DETAILED DESCRIPTION:
This proposal is in response to RFA-DA-04-008, Group Treatment for Individuals in Drug Abuse or Alcoholism Treatment. Of particular interest to the agencies are group therapies for Conduct Disordered adolescents, reducing the spread of infectious disease, and mechanisms of action. This proposal targets these areas of interest. This study will focus on treating substance abusing incarcerated teens using 2 individually administered Motivational Interviewing (MI) sessions followed by 10 group sessions of Cognitive Behavior Therapy (CBT). MI is conceptualized as preparation for group CBT. The control group receives individualized Relaxation Training (RT) followed by group Treatment as Usual (TU). Currently, t here is little research regarding effective group treatments for incarcerated teens and this study will address this gap in our knowledge base.

In this proposed randomized trial, a one-way design (MI/CBT vs RT/TU) will be used to determine whether MI/CBT enhances group therapy participation and reduces substance use and related problems (such as crime, injuries and unprotected sex) post discharge in substance-involved juvenile delinquents. RT/TU is based on the 12-step model and includes psycho-educational components. Participant are followed during incarceration and for 6 months post incarceration. Primary outcome variables include alcohol and marijuana use, as well as related behaviors (illegal activities, sex or injuries while drunk or high). It is hypothesized that in comparison to teens in RT/TU, youth receiving MI/CBT will participate more in therapy (according to teen, facility staff, and counselor ratings) and will show lower levels of substance use and related problems after discharge.

Frequently, substance abuse treatment is unavailable to youths in the juvenile justice system, and when treatment is available, it may be provided in group format using untested therapies. A motivation/skills-based intervention (delivered in group format) may prove efficacious in enhancing motivation and in reducing substance abuse and related problems. This study extends previous research by rigorously evaluating group treatment for incarcerated teens. We will examine processes contributing to the efficacy of group MI/CBT, and the influence of race and ethnicity on treatment effects. The development of effective interventions for substance using juvenile offenders has the potential to reduce substance abuse and crime in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents will be eligible if in the year prior to incarceration they either a) drank alcohol or used marijuana at least once per month or b) binge-drank (> 5 for boys, > 4 for girls) during any two week period; or they drank or used marijuana in the four weeks before the offense for which they were incarcerated; or they used alcohol or marijuana in the four weeks before they were incarcerated.

Exclusion Criteria:

Those teens sentenced for less than 4 months or greater than 12 months, those who are younger than 14 years or older than 19 years, and those for whom have inability to consent/assent (example, language barrier) are not obtained will be excluded from participation.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 205 (Actual)
Dates: Start 2004-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Stein, Ph.D., Principal Investigator — University of Rhode Island
Locations (1):
- Rhode Island Training School, Cranston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
With appropriate request and procedure.

REFERENCES:
- [Background] Martin RA, Stein LA, Clair M, Cancilliere MK, Hurlbut W, Rohsenow DJ. Adolescent Substance Treatment Engagement Questionnaire for Incarcerated Teens. J Subst Abuse Treat. 2015 Oct;57:49-56. doi: 10.1016/j.jsat.2015.04.011. Epub 2015 May 7. PMID 26021405
- [Background] Stein LA, Clair M, Martin RA, Soenksen S, Lebeau R, Rohsenow DJ, Kahler CW, Hurlbut W, Monti PM. Measuring behaviors of individual adolescents during group-based substance abuse intervention. Subst Abus. 2014;35(4):408-17. doi: 10.1080/08897077.2014.949337. PMID 25127289
- [Background] Bernstein MH, Stein LA. Do bisexual girls report higher rates of substance use than heterosexual girls? A failure to replicate with incarcerated and detained youth. J Bisex. 2015;15(4):498-508. doi: 10.1080/15299716.2015.1057889. Epub 2015 Nov 17. PMID 27087787
- [Background] Stein LA, Clair M, Rossi JS, Martin RA, Cancilliere MK, Clarke JG. Gender, ethnicity and race in incarcerated and detained youth: services and policy implications for girls. Psychiatr Rehabil J. 2015 Mar;38(1):65-73. doi: 10.1037/prj0000089. Epub 2014 Sep 1. PMID 25180525
- [Background] Stein LA, Clair M, Soenksen S, Martin RA, Clarke JG. Studying Process and Proximal Outcomes of Supervision for Motivational Interviewing. Train Educ Prof Psychol. 2015 May;9(2):175-182. doi: 10.1037/tep0000073. No abstract available. PMID 26417395
- [Background] Bassett SS, Stein LA, Rossi JS, Martin RA. Evaluating Measures of Fidelity for Substance Abuse Group Treatment With Incarcerated Adolescents. J Subst Abuse Treat. 2016 Jul;66:9-15. doi: 10.1016/j.jsat.2016.02.011. Epub 2016 Mar 9. PMID 27211991

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants withdrew or could not be located prior to treatment assignment.
Period: Overall Study
Arm/Group | MI/CBT | RT/TU
Started | 100 | 99
Completed | 79 | 84
Not Completed | 21 | 15
Not completed — Lost to Follow-up | 21 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MI/CBT | RT/TU | Total
Number analyzed (Participants) | 100 | 99 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.05 (1.01) | 17.11 (1.08) | 17.08 (1.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 88 | 91 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 47 | 79
  Not Hispanic or Latino | 68 | 52 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 9 | 16
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 42 | 39 | 81
  White | 33 | 37 | 70
  More than one race | 8 | 6 | 14
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 100 | 99 | 199

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use, Average # of Drinks Per Week
Description: using Time-Line Follow-back, we collected average # of drinks per week for a 3 month period at Baseline, 3 months and 6 months post release
Time Frame: Baseline, 3 months post release and 6 months post release
Population: Individuals dropped out of the project over time, more people were analyzed at Baseline than at each Follow-up assessment.
Measure: Mean (Standard Deviation); unit: average # of drinks per week
Arm/Group | MI/CBT | RT/TU
Number analyzed (Participants) | 100 | 98
average # of drinks per week
  Average # of drinks per week at Baseline | 11.16 (19.04) | 10.62 (17.02)
  Average # of drinks per week 3 months post release: number analyzed (Participants) | 82 | 89
  Average # of drinks per week 3 months post release | 5.16 (12.27) | 3.86 (9.16)
  Average # drinks per week at 6 months post release: number analyzed (Participants) | 79 | 84
  Average # drinks per week at 6 months post release | 7.08 (13.69) | 3.57 (7.57)

2. Primary Outcome: Marijuana Use
Description: using Time-Line Follow-back, we collected average number of joints per smoking day
Time Frame: Baseline, 3 months post release and 6 month post release
Population: Individuals dropped out of the study over time, more people were analyzed at baseline than at follow up assessments
Measure: Mean (Standard Deviation); unit: # of joints per smoking day
Arm/Group | MI/CBT | RT/TU
Number analyzed (Participants) | 100 | 98
# of joints per smoking day
  # of joints per smoking day at baseline | 5.84 (5.57) | 4.98 (4.25)
  # of joints per smoking day at 3 months: number analyzed (Participants) | 82 | 89
  # of joints per smoking day at 3 months | 2.52 (2.37) | 2.48 (2.49)
  # of joints per smoking day at 6 months: number analyzed (Participants) | 79 | 84
  # of joints per smoking day at 6 months | 2.48 (2.16) | 2.95 (3.71)

3. Primary Outcome: Crime: General Predatory Aggression
Description: using the Misbehaviors Questionnaire, we collect 12 items that assess the average number of times crimes involving predatory aggression were committed at Baseline, 3 months and 6 month post release.
Time Frame: Baseline, 3 months post release and 6 months post release
Population: Due to project drop out more people were analyzed at baseline than at both follow up assessments.
Measure: Mean (Standard Deviation); unit: Average # of times
Arm/Group | MI/CBT | RT/TU
Number analyzed (Participants) | 100 | 99
Average # of times
  6 month avg. # times of predatory aggression | 6.35 (3.72) | 1.92 (2.41)
  3 month post avg. # times of predatory aggression: number analyzed (Participants) | 82 | 89
  3 month post avg. # times of predatory aggression | 2.13 (2.69) | 1.92 (2.41)
  6 month post avg. # times of predatory aggression: number analyzed (Participants) | 79 | 84
  6 month post avg. # times of predatory aggression | 1.89 (2.71) | 1.44 (2.03)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were active on the study for 6 month period.
Arm/Group | MI/CBT | RT/TU
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 0/100 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes